## THE EFFECT OF MOTOR IMAGERY TRAINING ON MUSCLE ACTIVITY, MOTOR IMAGERY AND FUNCTIONAL MOVEMENT SKILLS IN INDIVIDUALS UNILATERAL CEREBRAL PALSY

**NCT NUMBER: 03954808** 

**Document Date: 10.06.2020** 

## **Study Protocol**

8 weeks, 2 sessions of with a 30 minutes physiotherapy training and 15 minutes motor imagery training, within a spesific program, was applied to motor imagery training group. 8 weeks, 2 sessions (45 minutes) of physiotherapy training was applied to Cerebral Palsy control group. The motor imagery training was applied one to one by the same specialist physiotherapist for all individuals with CP. Physiotherapy training; It consisted of physiotherapy training including weight transferring, strengthening and walking training. Evaluations made 3 times, before training, after training (8th week) and after training (14th week) for motor imagery and Cerebral Palsy control group. Typically developing individuals were evaluated once.